CLINICAL TRIAL: NCT05520840
Title: Evaluation of Peripheral Blood Protein Biomarkers for Colorectal Cancer Screening
Acronym: COLODIAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: OncoDiag (Unknown); University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/0149/HP
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
Keywords: biomarkers
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient referred for screening colonoscopy or for endoscopic resection (Experimental): Patient aged 50 years or older referred for screening colonoscopy after a positive fecal immunochemical test or for endoscopic resection of a previously identified suspicious colorectal lesion will have a blood sampling for biomarkers detection
  Interventions: Diagnostic Test: blood sampling for screening of biomarkers

INTERVENTIONS:
Diagnostic Test: blood sampling for screening of biomarkers — Patient aged 50 years or older referred for screening colonoscopy after a positive fecal immunochemical test or for endoscopic resection of a previously identified suspicious colorectal lesion will have a blood sampling for biomarkers detection

SUMMARY:
The aim of the study is to validate the value of value of peripheral blood protein biomarkers in colorectal cancer screening, and to identify new ones

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 years or older referred for screening colonoscopy after a positive FIT test or for endoscopic resection of a previously identified suspicious colorectal lesion

Exclusion Criteria:

* Very high risk of colorectal cancer: Lynch syndrome, Familial adenomatous polyposis, Peutz-Jeghers syndrome, Familial polyposis associated with a MutYH gene defect
* Other solid cancers or haematological malignancies that are progressive and/or undergoing treatment (apart from basal cell skin carcinoma)
* Contraindication to total colonoscopy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Number of patient with advanced neoplasia at colonoscopy | Day 1
Number of patient with presence of best isolated serum biomarkers selected from different candidates | Day 1

SECONDARY OUTCOMES:
Number of patient with presence of other isolated serum biomarkers selected from different candidates | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Grancher, MD, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - Clinique du Cèdre, Bois-Guillaume
  - Caen University Hospital, Caen
  - Dijon University Hospital, Dijon

IPD SHARING:
Plan to Share IPD: No